CLINICAL TRIAL: NCT04408391
Title: Descriptive Pilot Study of Brain MRI Imaging in Patients With SARS-Cov2 (COVID-19) Infection With or Without Anosmia
Brief Title: Brain MRI Imaging in Patients With SARS-Cov2 (COVID-19) Infection With or Without Anosmia
Acronym: ANOSIRM
Status: Withdrawn | Type: Observational
Why Stopped: No Inclusion potentiel
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2020-01/BL-001
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Covid-19; Anosmia
MeSH Terms: conditions — COVID-19; Anosmia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 patients with anosmia: Patients reporting loss of smell and scoring < 30 on a VAS 0-100 for ability to detect n-Butanol diluted 1/1000
  Interventions: Other: Brain MRI scan
- COVID-19 patients without anosmia: Patients reporting no loss of smell and scoring > 80 on a VAS 0-100 for ability to detect n-Butanol diluted 1/16000
  Interventions: Other: Brain MRI scan

INTERVENTIONS:
Other: Brain MRI scan — Resting state, functional, structural and morphometric MRI; diffusion tensor imaging on a 3-Tesla MRI scanner

SUMMARY:
To date there is no brain imaging and olfactory data available in COVID-19 positive patients with anosmia. By describing the pathophysiological characteristics underlying the olfactory symptoms and clinical characteristics of COVID-19 infection, the study investigators wish to compare the MRI aspects obtained in COVID-19 patients with and without anosmia, in the absence of other underlying neurological disorders.

DETAILED DESCRIPTION:
Brain mapping of COVID-19 patients with or without anosmia will allow better understanding of the mechanisms leading to the onset of these symptoms and will provide a pathophysiological basis for the therapeutic interventions to improve the clinical prognosis of affected patients.

The study investigators hypothesize that in COVID-19 patients witch anosmia the brain mapping objectified by an MRI examination is modified and that there are functional abnormalities in the brain in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients consulting the CAREB or hospitalized at the Nîmes teaching hospital due to COVID-19 infection (fever, persistent cough, tiredness, shortness of breath, diarrhea, abdominal pain, chest pain, sore throat, loss of smell or taste)
* COVID-19 confirmed by RT-PCR and / or chest CT or clinical characteristics (i.e an epidemic history and 2 clinical manifestations or at least 3 clinical manifestations)
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan "with anosmia" group:
* scoring < 30 on a VAS 0-100 for olfactory ability
* Responding "yes" to question "have you lost your sense of smell in the last few days?"
* Negative result to olfactory test with n-Butanol diluted to 1/1000. "without anosmia" group:
* scoring < 80 on a VAS 0-100 for olfactory ability
* Responding "no" to question "have you lost your sense of smell in the last few days?"
* Positive result to olfactory test with n-Butanol diluted to 1/16000.

Exclusion Criteria:

* Patient suffering from serious medical problems or hospitalized in an intensive care unit for invasive ventilation or severe dyspnea.
* Patient with neurological (motor, sensitive or cognitive), neuropsychiatric or vascular disorders.
* Patient with a contraindication to MRI (pace maker, claustrophobic patient, metallic heart valve, etc.).
* Patient with a history of rhinological pathology or a sense of smell problem.
* Patient with known neurological, psychiatric or neuroradiological manifestation.The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject is unable to express consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient is pregnant, parturient or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients consulting the CAREB or hospitalized at the Nîmes teaching hospital due to COVID-19 infection confirmed by RT-PCR and / or chest CT or clinical characteristics (i.e an epidemic history and 2 clinical manifestations or at least 3 clinical manifestations) with or without anosmia.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Brain regional homogeneity between COVID-19 patients with and without anosmia | Day 0
  MRI; Voxels

SECONDARY OUTCOMES:
Brain regional homogeneity between COVID-19 patients with and without anosmia | Month 3
  MRI; Voxels
Topography of supra- or sub-tentorial lesions between COVID-19 patients with and without anosmia | Day 0
  MRI; Voxels
Fractional anisotropy between COVID-19 patients with and without anosmia | Day 0
  MRI; voxels, value between 0-1
Fractional anisotropy between COVID-19 patients with and without anosmia | Month 3
  MRI; voxels, value between 0-1
Mean diffusivity between COVID-19 patients with and without anosmia | Day 0
  MRI; mm2/s
Mean diffusivity between COVID-19 patients with and without anosmia | Month 3
  MRI; mm2/s
Radial diffusivity between COVID-19 patients with and without anosmia | Day 0
  MRI; mm2/s
Radial diffusivity between COVID-19 patients with and without anosmia | Month 3
  MRI; mm2/s
Self-assessed olfactory and gustatory test | Day 0
  Four questions measured by 0-100 visual analogue scale: how do you rate the quality of your sense of smell/taste normally/today
Self-assessed olfactory and gustatory test | Day 8
  Four questions measured by 0-100 visual analogue scale: how do you rate the quality of your sense of smell/taste normally/today
Self-assessed olfactory and gustatory test | Month 1
  Four questions measured by 0-100 visual analogue scale: how do you rate the quality of your sense of smell/taste normally/today
Self-assessed olfactory and gustatory test | Month 2
  Four questions measured by 0-100 visual analogue scale: how do you rate the quality of your sense of smell/taste normally/today
Ability to detect odor | Day 0
  Ability to smell 1.5ml air freshner on a 0-100 VAS scale (cut-offs: strang (>80), moderate (40-80), attenuated (<40)
Ability to taste a pinch of sugar | Day 0
  Patient asked to describe whether a pinch of sugar on their tongue taste sweet or salty
Presence of thrombotic and hemorrhagic lesions | Day 0
  MRI: absence/presence
Presence of thrombotic and hemorrhagic lesions | Month 3
  MRI: absence/presence
Presence of lesions with hyperintensity | Day 0
  Short Ti Inversion Recovery (STIR); presence/absence
Presence of lesions with hyperintensity | Month 3
  Short Ti Inversion Recovery (STIR); presence/absence
Projection network analysis of all patients | Day 0
  beta voxels
Projection network analysis of all patients | Month 3
  beta voxels
Blinded independent component analysis of all patients | Day 0
  beta voxels
Blinded independent component analysis of all patients | Month 3
  beta voxels
default mode network analysis of all patients | Day 0
  beta voxels
default mode network analysis of all patients | Month 3
  beta voxels
executive control network analysis of all patients | Day 0
  beta voxels
executive control network analysis of all patients | Month 3
  beta voxels

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lallemant, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France